CLINICAL TRIAL: NCT05384795
Title: Perioperative Atelectasis in Patients Undergoing Orthopaedic Surgery: Prospective Cohort Study
Brief Title: Perioperative Atelectasis in Orthopaedic Surgery: a Prospective Study
Acronym: ATELHO
Status: Completed | Type: Observational
Sponsor: Eric Albrecht (Other)
Responsible Party: Sponsor-Investigator, Eric Albrecht, Prof. Dr. med, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Other Study IDs: CER-VD 2022-00712
Record Dates: First submitted 2022-05-13; First posted 2022-05-20 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General anesthesia
  Interventions: Other: Lung ultrasound
- Spinal anesthesia
  Interventions: Other: Lung ultrasound
- Peripheral nerve block
  Interventions: Other: Lung ultrasound

INTERVENTIONS:
Other: Lung ultrasound — Lung atelectasis score

SUMMARY:
This study aims at comparing a perioperative pulmonary atelectasis score, measured by pulmonary ultrasound, in patients operated undergoing orthopedic surgery under general anesthesia, spinal anesthesia or peripheral nerve block. The association between the atelectasis score and previously identified risk factors will be studied.

DETAILED DESCRIPTION:
Atelectasis is one of the most common pulmonary complications in the perioperative period, occurring in 85% to 90% of patients under general anesthesia. It can be responsible for hypoxemia and be associated with postoperative pulmonary complications such as pneumonia. The consequences are a prolongation of the hospital stay and an increase in mortality.

The appearance of perioperative atelectasis is mainly secondary to the induction of general anesthesia with an incidence up to 90%. The different causes are, for example, the administration of muscle relaxants, mechanical ventilation and the position of the patient.

In orthopedic surgery, many procedures are performed under spinal anesthesia or under peripheral nerve block. At present, there are no studies measuring the incidence of atelectasis in patients operated under these two techniques of locoregional anesthesia, with the exception of parturients undergoing cesarean section.

This study aims at comparing a perioperative pulmonary atelectasis score, measured by pulmonary ultrasound, in patients operated undergoing orthopedic surgery under general anesthesia, spinal anesthesia or peripheral nerve block. The association between the atelectasis score and previously identified risk factors will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18;
* Patients scheduled for an elective operation at the Orthopedic Hospital of CHUV;
* Signature of the study consent

Exclusion Criteria:

* Thoracic deformities preventing the performance of pulmonary ultrasound (dressings, drains, fractures, etc.);
* Refusal to participate;
* Patient does not speak French.
* Inability to discern

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be patients scheduled for elective surgery at the Orthopedic Hospital from CHUV.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Lung atelectasis score | immediately after the surgery
  Atelectasis score based on validated ultrasound quantification (comparing different anesthesia techniques)

SECONDARY OUTCOMES:
Lung atelectasis score | Four timepoints: at baseline, immediatly before surgery (after anesthesia induction), immediately after the surgery, and at the recovery room
  Atelectasis score

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Fully anonymised IPD will be shared upon reasonable request.